CLINICAL TRIAL: NCT01155037
Title: Phase 2 Study to Evaluate the Safety of and the Immunogenicity to an Adjuvanted A(H1N1)v Influenza Vaccine in HIV-Infected Adults
Brief Title: Safety of and Immunogenicity to an H1N1 Influenza Vaccine in HIV-infected Adults
Acronym: VIP-H1N1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Marilia Santini de Oliveira, Medical doctor, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VIP-H1N1
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: HIV Infection
Keywords: HIV, influenza A H1N1, vaccine
MeSH Terms: conditions — HIV Infections; Orthomyxoviridae Infections | interventions — halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3.75 µg of the vaccine on days 0 and 21 (Experimental): Patients infected with HIV will receive 3.75 µg of an adjuvanted A H1N1 vaccine in two applications 21 days apart.
  Interventions: Biological: Adjuvanted vaccine against H1N1 influenza virus (GSK)
- 7.5 µg of the vaccine on days 0 and 21 (Experimental): Patients infected with HIV will receive 7.5µg of an adjuvanted A H1N1 vaccine in two applications 21 days apart.
  Interventions: Biological: Adjuvanted vaccine against H1N1 influenza virus (GSK)
- 3.75 µg of the vaccine on day 0 (Active Comparator): The volunteers in the control group will receive a single application of 3.75 µg dose of the vaccine.
  Interventions: Biological: Adjuvanted vaccine against H1N1 influenza virus (GSK)

INTERVENTIONS:
Biological: Adjuvanted vaccine against H1N1 influenza virus (GSK) — Patients infected with HIV will receive 3.75 µg of an adjuvanted A H1N1 vaccine in two applications 21 days apart.
  Arms: 3.75 µg of the vaccine on days 0 and 21
Biological: Adjuvanted vaccine against H1N1 influenza virus (GSK) — Patients infected with HIV will receive 7.5 µg of an adjuvanted A H1N1 vaccine in two applications 21 days apart.
  Arms: 7.5 µg of the vaccine on days 0 and 21
Biological: Adjuvanted vaccine against H1N1 influenza virus (GSK) — Control group will receive 3.75 µg of an adjuvanted A H1N1 vaccine in one single application.
  Arms: 3.75 µg of the vaccine on day 0

SUMMARY:
This is a randomized, open label, phase II trial to evaluate the safety and immunogenicity of two different schedules of vaccination against influenza A H1N1 in HIV-infected individuals, in which each of the randomized groups will be compared with HIV-negative volunteers vaccinated with the regimen indicated by the Brazilian National Immunization Program. Will be included in the study HIV-infected patients, stratified by CD4 count (< 200 cells/mm3 or > 200 cells/mm3) at the time of screening for the study, not receiving antiretroviral therapy treatment or receiving stable treatment for at least 8 weeks, with no plans to change over the next 6 months, eligible to receive vaccine against influenza A H1N1. The control group will be formed by HIV-negative individuals, confirmed by serology performed at screening, eligible to receive vaccine against influenza A H1N1. Patients infected with HIV will receive one of two possible vaccination regimens: 1) 3.75 µg in two applications 21 days apart, 2) 7.5 µg in two applications 21 days apart. The volunteers in the control group will receive a single application of 3.75 µg dose of the vaccine. The study's hypotheses are: 1) The vaccine against the H1N1 virus promotes antibody titers above the level specified for protection (seroconversion), being as safe and well tolerated in patients HIV-1 infected as in non HIV-infected volunteers; 2) The proportion of seroconversion for H1N1 virus vaccine at a dose of 3.75 µg in HIV-1-infected patients is similar to the proportion of seroconversion induced by the same vaccine at a dose of 7.5 µg; 3)The proportion of seroconversion with one dose of the vaccine against H1N1 virus is similar to the proportion after the second dose.

ELIGIBILITY:
Inclusion Criteria - for all participants

* Both genders, aged between 18 and 59 years;
* Capacity to give informed consent voluntarily to participate in the study;
* Study participants with reproductive potential (defined as girls after menarche or women who have not reached menopause at least during 24 consecutive months, or who menstruated during the past 24 months, or have not undergone surgical sterilization) must have pregnancy test negative results, in blood or urine, at screening and in the vaccine application days. If they have sexual practices likely to promote pregnancy, the participants must use some form of contraception during the study period. At least one of the following methods MUST be properly used: Condoms (male or female, Hormonal contraceptive.
* Laboratory results in the study screening: hemoglobin > 8.0 g/dL; Direct bilirubin < 2.5 x the upper limit of normal; Alanine aminotransferase, ALT (SGPT) and aspartate aminotransferase, AST (SGOT) < 3 x the upper limit of normal; Platelet count > 100.000/mm3

Inclusion Criteria - unique to the participants with HIV infection:

* HIV-1 infection (as evidenced by rapid HIV testing or ELISA kit approved and confirmed by repeating the ELISA, IFA, Western blot, HIV-1 plasma viral load) at any time before entering the study.
* Without changing the antiretroviral treatment within 8 weeks prior to the screening for the study: If the volunteer is receiving HAART he/she is required to be using the same regimen within at least 8 weeks before screening. Changes in antiretroviral dosage within 8 weeks prior to entering the study are permitted. In addition, the exchange of pharmacological formulation (eg. the conventional formulation for combination formulations) is allowed. If the volunteer is not on regular antiretroviral treatment, he/she should not have received any dose of any antiretroviral within 8 weeks prior to screening, including for the prevention of HIV vertical transmission (previous prophylactic and therapeutic regimens are allowed)
* Without planning to change or start HAART in the next 6 months.

Inclusion criteria - unique to the participants without HIV infection (control group):

* HIV-negative test result documented by rapid test approved in Brazil
* Health professionals with indication of receiving H1N1 virus vaccine

Exclusion Criteria:

* Use of any systemic anticancer or immunomodulator treatment, corticosteroid, experimental vaccines, interleukins, interferons, growth factors or intravenous immunoglobulin (IVIG) within 45 days prior to entry into the study.
* Pregnancy or lactation.
* Allergy and/or sensitivity or any known hypersensitivity to residues present in the vaccine (egg, chicken protein, egg albumin, formaldehyde, gentamicin sulphate and sodium deoxycholate) and/or thimerosal.
* Use of alcohol or addiction or other conditions which in the opinion of the site's investigator, may interfere with compliance to the study requirements.

D5. Serious illness requiring systemic treatment and/or hospitalization within 45 days prior to entry into the study

* Severe febrile illness or acute infection at the time of screening for the study and/or days of vaccination
* Vaccination against seasonal influenza in the last 12 months prior to study entry
* Previous vaccination against influenza A H1N1
* History or family history of Guillain-Barré Syndrome (parents, siblings, half-siblings or children).
* Diagnosis of neurological condition including (but not limited to) the absence of deep tendon reflexes, Achilles and patellar, in both legs (four missing) in the last six months.
* Disproportionate force loss in lower limb(s) compared to the upper limbs in the last six months.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
proportions of seroconversion | 21 days after vaccination regimen
  proportions of seroconversion for influenza A H1N1 in each of the four subsets of HIV-positive patients, and in the control group
proportions of seroprotection | 21 days after vaccination regimen
  proportions of seroprotection for influenza A H1N1 in each of the four subsets of HIV-positive patients and in the control group
Safety of the A H1N1 vaccine at two different regimens in HIV-infected adults | 1 months after vaccination
  Safety and tolerability of the vaccine against H1N1 virus in different doses and administration regimens in IV-infected adults

SECONDARY OUTCOMES:
Prevalence of A H1N1 influenza symptomatic disease in the study population | 12 months after vaccination
  proportions of the vaccine's protective factor against influenza A H1N1 in each of the four subsets of HIV-positive patients and in the control group
Persistence of antibodies against H1N1 virus | 12 months after vaccination
  Evaluate the persistence of antibody titers against H1N1 virus after the vaccine series in HIV-infected patients and control group
Changes in HIV viral load and CD4 | 12 months after vaccination
  Assess changes in HIV-1 viral load and CD4+ counts after the vaccine series.
Cellular immune responses to H1N1 vaccination in HIV-infected patients | 12 months after vaccination
  Determine the cellular immune responses and their correlation to the development and magnitude of responses to H1N1 virus, and compare the cellular immune responses

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) - Fiocruz, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Santini-Oliveira M, Camacho LA, Souza TM, Luz PM, Vasconcellos MT, Giacoia-Gripp CB, Morgado MG, Nunes EP, Lemos AS, Ferreira AC, Moreira RI, Veloso VG, Siqueira MM, Grinsztejn B. H1N1pdm09 adjuvanted vaccination in HIV-infected adults: a randomized trial of two single versus two double doses. PLoS One. 2012;7(6):e39310. doi: 10.1371/journal.pone.0039310. Epub 2012 Jun 25. PMID 22761759